CLINICAL TRIAL: NCT04583839
Title: SWEET: Sustaining Women's Engagement and Enabling Transitions After Gestational Diabetes Mellitus
Brief Title: SWEET: Postpartum Navigation After GDM
Acronym: SWEET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Lynn M Yee, Assistant Professor, Division of Maternal-Fetal Medicine Department of Obstetrics and Gynecology, Northwestern University, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00212306; 1R34DK125958 (NIH)
Record Dates: First submitted 2020-09-29; First posted 2020-10-12 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Gestational Diabetes; Preventive Care / Anticipatory Guidance; Retention in Care; Postpartum Health; Lifestyle Modification
MeSH Terms: conditions — Diabetes, Gestational | interventions — Patient Navigation

STUDY DESIGN:
Intervention Model Description: There will be two cohorts. One cohort will be provided intensive, individualized patient navigation services through one year postpartum, with a focus on diabetes prevention. The second cohort will receive usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Navigation Group (Experimental): Women who are randomized into SWEET will be assigned to a patient navigator. The navigator will meet women during hospitalization, at postpartum appointments, during primary care appointments, and as needed. At these face-to-face meetings, the navigator will perform education about the postpartum OGTT, post-GDM management plan, diabetes mellitus risks, lifestyle modification, and primary care transition. The navigator will facilitate the development of an individualized GDM Care Plan in conjunction with the patient and the medical team. The navigator will assess individual barriers to T2DM screening and prevention. At appointments, the navigator will also ensure a woman understands her diabetes-related care plan and will perform health education and barrier-reducing tasks as needed.
  Interventions: Behavioral: Patient Navigation Program
- Non-navigation cohort (No Intervention): No navigation will be provided; women will receive usual care.

INTERVENTIONS:
Behavioral: Patient Navigation Program — SWEET is a GDM-focused intervention that will apply barrier-reduction patient navigation strategies to improve health after a pregnancy with GDM. Women in SWEET will receive GDM-specific, tapered, individualized navigation services, including logistical support, psychosocial support, and patient education, through 1-year postpartum.
  Other Names: SWEET
  Arms: Navigation Group

SUMMARY:
This study is a pilot assessment of Sustaining Women's Engagement and Enabling Transitions after GDM (SWEET), a GDM-focused intervention that will apply barrier-reduction patient navigation strategies to improve health after a pregnancy with gestational diabetes mellitus. The investigators aim to determine, via a randomized controlled trial of 40 women who have had GDM, whether those who receive the navigation intervention have improved diabetes-related health at 1 year after birth compared to those who receive usual care. The SWEET intervention will provide GDM-specific, individualized navigation services that leverage existing clinical infrastructure, including logistical support, psychosocial support, and health education, through 1-year postpartum. Participants will undergo surveys, interviews, and medical record review at multiple time points. The investigators will also conduct qualitative interviews with clinical providers.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) poses a substantial long-term health burden to women due to the 7-fold increased risk of developing type 2 diabetes mellitus (T2DM) and other cardiovascular disorders. Yet, there are many gaps in the transition period after GDM, which is a particularly critical time due to enhanced motivation and access. Nevertheless, a minority of women receive postpartum screening for dysglycemia or have successful transition to primary care. Although T2DM prevention interventions can be successful, they cannot be deployed without retention and engagement in care. Addressing the unique barriers experienced by postpartum women requires innovative models of health care delivery to promote prevention of T2DM after GDM. One potential intervention with demonstrated successes in other arenas is patient navigation, a barrier-focused, longitudinal, patient-centered intervention that offers support for a defined set of health services.

This protocol is to perform a pilot assessment of Sustaining Women's Engagement and Enabling Transitions after GDM (SWEET), a GDM-focused intervention that will apply barrier-reduction patient navigation strategies to improve health after a pregnancy with GDM. The investigators aim to determine, via a randomized controlled trial of 40 women who have had GDM, whether those who receive the SWEET navigation intervention have improved diabetes-related health at 1 year after birth compared to those who receive usual care. In order to promote self-efficacy, enhance access, and sustain long-term engagement, the SWEET intervention will provide GDM-specific, individualized navigation services that leverage existing clinical infrastructure, including logistical support, psychosocial support, and health education, through 1-year postpartum.

Aim 1 will evaluate whether clinical (weight, glycemic control, abdominal circumference, and blood pressure), health services (postpartum and primary care visit attendance), and patient-reported (diabetes self-efficacy, activation, and T2DM risk perception) outcomes differ in women exposed to SWEET versus usual care. Aim 2 will evaluate feasibility and acceptability. This proposal will generate key data for the conduct of a full-scale trial of a GDM-specific postpartum patient navigation program that will address critical questions about long-term maternal health and T2DM prevention.

SWEET bridges the chasm between care during pregnancy - focused on improving the health of the pregnant woman and her offspring - and long-term women's health care - focused on chronic disease management and preventive health. The long-term goals are to understand how to optimize long-term health after GDM in order to prevent or ameliorate the effects of T2DM beyond the perinatal period.

ELIGIBILITY:
Patient Participants:

Inclusion Criteria:

* Pregnancy delivering at or after 30 weeks of gestation, regardless of neonatal outcome
* Gestational diabetes mellitus, treatment of any modality
* English- or Spanish- speaker
* Age 16 or greater
* Established patient at the Northwestern Medicine obstetrics and gynecology practices

Exclusion Criteria:

* Intent to transfer prenatal care to an outside institution or leave Chicago region
* Pre-gestational diabetes mellitus
* Weight loss during pregnancy
* History of bariatric surgery
* Prior enrollment in SWEET
* Enrollment in a concurrent research study that poses a potential conflict to the aims of SWEET or the other study

Health care provider participants:

Inclusion Criteria:

* Age 18 or greater
* English-speaking
* Obstetrician or advanced practitioner who has provided postpartum care to a participating SWEET participant OR primary care provider who has provided primary care to a participating SWEET participant

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Postpartum weight retention | 1 year postpartum
  Difference between 1) preconception weight and 2) weight at 1 year postpartum,

SECONDARY OUTCOMES:
Postpartum diabetes screening completion | 4-12 weeks postpartum
  Number of women with completion of a 2-hour oral glucose tolerance test by 12 weeks postpartum.
Postpartum diabetes screening result | 4-12 weeks postpartum
  Result of postpartum OGTT.
Abdominal circumference | 4-12 weeks and 1 year postpartum
  Abdominal circumference at any time point in the first year after giving birth.
Blood pressure | 4-12 weeks and 1 year postpartum
  Blood pressure at any time point in the first year after giving birth and proportion with hypertension.
Postpartum visit attendance | 4-12 weeks postpartum
  Attendance at a comprehensive postpartum care visit by 12 weeks postpartum.
Assessment of postpartum glycemic control | 1 year postpartum
  Number of women who complete any measure of glycemic control (fasting glucose, random glucose, and/or hemoglobin A1c) by 1 year postpartum.
Postpartum transition to primary care | 1 year postpartum
  Number of women with appointment made and kept for primary care by 1 year postpartum.
Diabetes self-efficacy | 4-12 weeks and 1 year postpartum
  Diabetes Empowerment Scale (DES)- Minimum score is 1, and maximum score is 5. Higher scores indicate greater levels of diabetes self-efficacy.
Patient activation | 4-12 weeks and 1 year postpartum
  Patient Activation Measure (PAM)- Patient knowledge, skill, and confidence for managing one's own health and healthcare. Minimum score is 1, and maximum score is 100. Higher scores indicate higher activation levels in self-management.
Diabetes risk perception | 4-12 weeks and 1 year postpartum
  Risk Perception Survey for Developing Diabetes (RPS-DD)- adapted for women with gestational diabetes- Scores are averaged with higher scores indicating a greater personal control to prevent development of DM. Minimum score of 1, and maximum score of 5. Higher scores indicate greater personal control beliefs.

OTHER OUTCOMES:
Participant experiences and perspectives on GDM | 4-12 weeks and 1 year postpartum
  Qualitative feedback on experience with the GDM diagnosis, barriers to obtaining postpartum GDM-related care, and barriers and facilitators of the primary care transition.
Patient experiences with navigation | 4-12 weeks and 1 year postpartum
  Participants who are randomized to receive navigation will complete in-depth interviews about experiences with the program and areas for improvement.
Health care providers experiences with SWEET | Through completion of study, an average of 2 years
  Health care providers whose patients participate in the trial will undergo in-depth interviews about provider perceptions of the program, barriers to providing optimal care for women who have had GDM, the methods by which providers and the health care system can adopt postpartum care recommendations, and how to optimize SWEET for future study.
Patient satisfaction with logistical aspects of navigation | 4-12 weeks and 1 year postpartum
  Patient Satisfaction with Logistical Aspects of Navigation (PSN-L)- Participants randomized to navigation will complete surveys designed to understand their logistical experiences with patient navigation. Minimum score is 0, and maximum score is 78. Higher scores indicate higher levels of satisfaction.
Patient satisfaction with interpersonal relationship with navigator | 4-12 weeks and 1 year postpartum
  Patient Satisfaction with Interpersonal Relationship with Navigator (PSN-I)- Participants randomized to navigation will complete surveys designed to understand their interpersonal experiences with patient navigation. Minimum score is 0, and maximum score is 45. Higher scores indicate higher levels of satisfaction.
Proportion of eligible participants who enroll | Through completion of study, an average of 2 years
  Proportion of eligible participants who enroll will be defined as the proportion of women who enroll out of all approached, eligible women.
Recruitment rate | Through completion of study, an average of 2 years
  Recruitment rate will be defined as the number of women successfully enrolled per week during the study, using mean or median to illustrate the variation of the numbers.
Time to enrollment | Through completion of study, an average of 2 years
  Time to enrollment will be defined as the number of months to enroll target sample size.
Dropout rate | Through completion of study, an average of 2 years
  Dropout rate will be defined as the number of enrolled women who drop out of study participation during the 1-year follow-up per week.
Retention rate | Through completion of study, an average of 2 years
  Retention rate will be defined as the proportion of enrolled women who successfully complete all study visits during 1-year follow-up period.
Participant adherence with navigation | Through completion of study, an average of 2 years
  The participant adherence (engagement rate) outcomes will be calculated both as a proportion (percent of navigator-attempted contacts with response) and count (number of navigator-attempted contacts with response) among participants randomized to navigation. Feasibility targets will be defined as 80% recruitment, retention, and adherence rates. Targets are set at 80% based on prior literature using this threshold to represent greater engagement.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn M Yee, MD, MPH, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No